CLINICAL TRIAL: NCT02620384
Title: Metolazone As Early Add On Therapy For Acute Decompensated Heart Failure (MELT-HF)--A Single Center Pilot Study.
Acronym: MELT-HF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Limited resources available to met accrual goal.
Sponsor: Aultman Health Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015.03.26.F2
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Metolazone; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Placebo (Placebo Comparator): This group will receive all standard heart failure therapy and placebo pill.
  Interventions: Drug: Experimental: Placebo
- Experimental: Metolazone (Active Comparator): This group will receive all standard heart failure therapy with addition of metolazone.
  Interventions: Drug: Experimental: Metolazone

INTERVENTIONS:
Drug: Experimental: Placebo — All patients will receive standard heart failure therapy, including but not restricted to diuretics, digoxin, angiotensin converting enzyme inhibitors or angiotensin II receptor blockers, beta blockers, aldosterone antagonists, hydralazine, and/or nitrates, at the discretion of the treating physician. After informed consent is obtained, patients will be randomized 1:1 to the treatment arm or placebo arm. The first placebo dose is given within six hours of admininstration of first dose of intravenous diuretic. The second placebo dose is given at 24-hours after the first dose.
  Arms: Experimental: Placebo
Drug: Experimental: Metolazone — All patients will receive standard heart failure therapy, including but not restricted to diuretics, digoxin, angiotensin converting enzyme inhibitors or angiotensin II receptor blockers, beta blockers, aldosterone antagonists, hydralazine, and/or nitrates, at the discretion of the treating physician. After informed consent is obtained, patients will be randomized 1:1 to the treatment arm or placebo arm. The first dose of metolazone is given within six hours of admininstration of first dose of intravenous diuretic The second dose of metolazone is given 24-hours after the first dose.
  Arms: Experimental: Metolazone

SUMMARY:
The primary objective of the study is to determine efficacy of metolazone as synergistic therapy with Lasix in patients with acute decompensated heart failure. This will be a single center double blinded randomized placebo- controlled pilot study of the addition of 5 mg of metolazone per day for 2 days compared to placebo in patients admitted with acute decompensated heart failure.

DETAILED DESCRIPTION:
Heart failure is a major source of morbidity, mortality and growing public health cost. In US, the number of congestive heart failure patients is more than 4 million with more than 550,000 new annually reported cases. The annual cost of heart failure management exceeds 35 billion dollars per year.The heart failure readmissions and average length of hospital stay cost approximately $11,000 per patient.

Loop diuretics are used alone in the majority of cases to promote diuresis. An association of increased creatinine and increased risk of renal dysfunction, the cardiorenal syndrome, in the face of high dose loop diuretics has raised questions regarding the safety and toxicity of high dose loop diuretics. While the dose of diuretics is ubiquitous, little data exists to guide their use and many clinicians are uncertain as to when and how to initiate and limit therapy.

Prospective randomized data on large number of decompensated heart failure patients receiving metolazone in addition to standard therapy is scarce and needs further definitive evaluation in terms of clinical outcomes and safety. In many cases, a "stepped approach" with oral loop diuretics advancing to intravenous and finally combination high dose diuretics is employed.

Primary endpoint: Total urinary output and negative fluid balance in millilitres (ml) at 48 hours following first dose of intravenous diuretic.

Secondary endpoints:

1. Change in weight from admission to day 2.
2. Degree of improvement in dyspnea at 6,12, 24,36, and 48 hours assessed with Modified Borg Scale (1-10)
3. All cause mortality at 30 days.

This is a single center study of at least 200 patients who are admitted to Aultman Hospital with clinical decompensated congestive heart failure ( NYHA III-IV). It is a double blinded randomized placebo- controlled pilot study of the addition of 5 mg of metolazone per day for 2 days compared to placebo in patients admitted with acute decompensated heart failure. We will compare a strategy of early institution of metolazone with standard of care in patients admitted with decompensated heart failure and volume overload. All patients will receive standard heart failure therapy, including but not restricted to diuretics, digoxin, angiotensin converting enzyme inhibitors or angiotensin II receptor blockers, beta blockers, aldosterone antagonists, hydralazine, and/or nitrates, at the discretion of the treating physician.

After informed consent is obtained, patients will be randomized 1:1 to the treatment arm or placebo arm. Two additional doses of metolazone within 6 and 24 hours of administration of standard intravenous diuretics will be given to the treatment arm. Patients and physicians will be blinded to the administered drug (metolazone vs placebo).Drug will be distributed by pharmacy when a patient is consented and enrolled in the trial. Specific guidance/recommendations regarding diuretic therapy will be provided (documented in detail below) but will be at the discretion of the treating physician. We will collect data on demographics, co-morbidities, clinical presentations and outcomes with metolazone administration with patient follow up at one week (+3) and 30 (±7) days post discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Current hospitalization for chronic congestive heart failure with admission up to 48 hours prior to inclusion.
* Chronic heart failure will be defined as requiring treatment for a minimum of 30 days prior to current admission, NYHA Class III or IV at the time of hospitalization, and left ventricular ejection fraction less than 40% within one year or evidence of heart failure with preserved ejection fraction and evidence of diastolic dysfunction on echocardiogram.
* Admitted with clinical decompensated heart failure based on history, physical exam, and parameters indicating extracellular volume expansion such as including JVP ≥ 8 cm of water and 1+ or greater peripheral edema
* Is able to be dosed with study medication within six (6) hours of first dose of IV diuretics

Exclusion Criteria:

* Baseline severe hypotension (Mean arterial pressure < 55 mm Hg)
* Creatinine clearance less than 20 ml/min or creatinine greater than 2.5 mg/dl.
* Serum sodium less than 128 meq/L.
* Serum Potassium < 3.0 meq/L.
* Known adverse reaction to metolazone
* Inability to take oral medications
* Severe Aortic Stenosis (AVA < 0.8cm2)
* History of Hypertrophic obstructive cardiomyopathy
* Metastatic Carcinoma per history
* Severe COPD, FEV < 1L
* Severe dyspnea requiring prolonged CPAP,BIPAP or intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Chaudhry, MD, Principal Investigator — Aultman Health Foundation
Locations (1):
- Aultman Health Foundation, Canton, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 147 participants from one local institution (inpatient hospital) were enrolled between October 2015 and November 2017
Pre-assignment Details: Participants who signed consent but after further evaluation did not to meet inclusion or met one or more exclusion criteria were not included in the analysis. There were four screen failures following consent.
Period: Overall Study
Arm/Group | Experimental: Placebo | Experimental: Metolazone
Started | 70 | 73
Completed | 66 (Per protocol design patients must receive both doses of investigational product to be in analysis.) | 66 (Per protocol design patients must receive both doses of investigational product to be in analysis.)
Not Completed | 4 | 7
Not completed — Adverse Event | 2 | 1
Not completed — Discharged prior to 2nd dose | 2 | 5
Not completed — Drug shortage prevented 2nd dose | 0 | 1

BASELINE CHARACTERISTICS:
Population: Per protocol only participants who receive both doses of investigational product are analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Placebo | Experimental: Metolazone | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.67 (13.5) | 71.86 (12.8) | 72.77 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 40 | 37 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 63 | 64 | 127
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 66 | 66 | 132
NYHA Class at Enrollment [Number; unit: participants] — Class I: Patients with cardiac disease but no limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain.
  Class II (Mild) Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in above symptoms Class III (Moderate) Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes above symptoms.
  Class IV (Severe) Inability to carry on any physical activity without symptoms, may be present at rest.
  participants
    Class 3 | 28 | 25 | 53
    Class 4 | 38 | 41 | 79
N-Terminal proBNP Value Upon Admission [Mean (Standard Deviation); unit: pg/mL] | 10905.6 (12749.9) | 10184.7 (11340.1) | 10545.12 (12024.2)
Time Difference Qualifying Diuretic and Study Drug Initiation [Mean (Standard Deviation); unit: minutes] — Time difference between the first diuretic administered following presentation (Qualifying Diuretic) and the first dose of Study Drug
  minutes | 147.7 (147.7) | 121.3 (112.9) | 132.5 (114.3)

OUTCOME MEASURES:

1. Primary Outcome: Total Urinary Output at 48 Hours
Description: Total urinary output in milliliters (ml) at 48 hours. Measurement timing began with administration of first dose of investigational product, ended 48 hours later.
Time Frame: 48 hours
Population: All participants who received both doses of the investigational product and completed the 48 hour assessments were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Experimental: Placebo | Experimental: Metolazone
Number analyzed (Participants) | 66 | 66
Milliliters | 6893.777 (3122.6532) | 9333.288 (4188.5731)
Statistical Analysis 1: Comparison: Experimental: Placebo vs Experimental: Metolazone; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 2439.5110, 95% CI 2-sided [1160.8485 to 3718.1734], Standard Error of Mean 646.2707

2. Primary Outcome: Fluid Balance at 48 Hours
Description: Difference in value between input and output in milliliters (ml) at 48 hours. Measurement timing began with administration of first dose of investigational product, ended 48 hours later. Fluid balance = Fluid in minus Fluid out.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Mililiters
Arm/Group | Experimental: Placebo | Experimental: Metolazone
Number analyzed (Participants) | 66 | 66
Mililiters | -4260.762 (2705.8710) | -6510.091 (4121.3808)
Statistical Analysis 1: Comparison: Experimental: Placebo vs Experimental: Metolazone; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -2249.3294, 95% CI 2-sided [-3454.4999 to -1044.1589], Standard Error of Mean 608.2782

3. Secondary Outcome: Change in Weight First 48 Hours
Description: Change in weight from the date/time of study enrollment (baseline) and 48 hours.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: killograms
Arm/Group | Experimental: Placebo | Experimental: Metolazone
Number analyzed (Participants) | 66 | 66
killograms | -3.23227 (2.538462) | -5.93939 (4.033661)
Statistical Analysis 1: Comparison: Experimental: Placebo vs Experimental: Metolazone; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -2.717121, 95% CI 2-sided [-3.8637732 to -1.546510], Standard Error of Mean .586647

4. Secondary Outcome: Degree of Improvement in Dyspnea at 6, 12, 24, 36 and 48 Hours.
Description: Dyspnea assessed at 6, 12, 24, 36 and 48 hours with Modified Borg Scale (1-10). Range is from 1 (very slight) to 10 (maximal) dyspnea.
Time Frame: 6, 12, 24, 36 and 48 hours.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Placebo | Experimental: Metolazone
Number analyzed (Participants) | 66 | 65
score on a scale
  Baseline | 9 (.0000) | 9 (.0000)
  6 hours | 6.21 (1.524) | 5.49 (1.532)
  12 hours | 4.88 (1.564) | 3.98 (1.441)
  24 hours | 3.77 (1.662) | 2.95 (1.643)
  36 hours | 2.924 (1.6249) | 2.123 (1.5663)
  48 hours | 2.295 (1.6640) | 1.600 (1.5441)
Statistical Analysis 1: Comparison: Experimental: Placebo vs Experimental: Metolazone; Test type: Superiority; p = .014, t-test, 2 sided — Represents BORG_48_hours; Mean Difference (Final Values) = -.6955, 95% CI 2-sided [-1.2506 to -.1403], Standard Error of Mean .2806 — Method of estimation is for 48 hour measure

5. Secondary Outcome: Total Dose Diuretics First 48 Hours
Description: Total dosage loop diuretic in first 48 hours using conversion tool to calculate intravenous Lasix equivalence
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Experimental: Placebo | Experimental: Metolazone
Number analyzed (Participants) | 66 | 65
Milligrams | 346.470 (381.9480) | 350.160 (444.8640)
Statistical Analysis 1: Comparison: Experimental: Placebo vs Experimental: Metolazone; Test type: Superiority; p = .959, t-test, 2 sided; Mean Difference (Final Values) = 3.6903, 95% CI 2-sided [-1395694 to 147.1545], Standard Error of Mean 72.4074

6. Secondary Outcome: Number of Participants With Inotrope Administration During First 48 Hours
Description: Number of Participants with Inotrope administration during first 48 hours following study enrollment.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Placebo | Experimental: Metolazone
Number analyzed (Participants) | 66 | 66
Participants | 9 | 4
Statistical Analysis 1: Comparison: Experimental: Placebo vs Experimental: Metolazone; Test type: Superiority; p = .144, Chi-squared

7. Secondary Outcome: All Cause Mortality at 30 Days
Description: All Cause Mortality at 30 Days
Time Frame: 30 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Placebo | Experimental: Metolazone
Number analyzed (Participants) | 66 | 66
Participants | 1 | 4
Statistical Analysis 1: Comparison: Experimental: Placebo vs Experimental: Metolazone; Test type: Superiority; p = .171, Chi-squared

8. Other Pre Specified Outcome: Length of Hospital Stay
Description: Length of hospital stay in days
Time Frame: Inpatient Hospitalization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Experimental: Placebo | Experimental: Metolazone
Number analyzed (Participants) | 66 | 66
days | 5.33 (4.695) | 5.44 (3.672)
Statistical Analysis 1: Comparison: Experimental: Placebo vs Experimental: Metolazone; Test type: Superiority; p = .885, t-test, 2 sided; Mean Difference (Final Values) = .106, 95% CI 2-sided [-1.346 to 1.558], Standard Error of Mean .734

9. Other Pre Specified Outcome: All Cause Readmission Within 30 Days
Description: All Cause Readmission Within 30 Days
Time Frame: 30 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Placebo | Experimental: Metolazone
Number analyzed (Participants) | 66 | 66
Participants | 10 | 9
Statistical Analysis 1: Comparison: Experimental: Placebo vs Experimental: Metolazone; Test type: Superiority; p = .804, Chi-squared

10. Other Pre Specified Outcome: Heart Failure Readmission Within 30 Days
Description: Heart Failure Readmission Within 30 Days
Time Frame: 30 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Placebo | Experimental: Metolazone
Number analyzed (Participants) | 66 | 66
Participants | 2 | 4
Statistical Analysis 1: Comparison: Experimental: Placebo vs Experimental: Metolazone; Test type: Superiority; p = .403, Chi-squared

11. Other Pre Specified Outcome: Number of Participants With Potassium Electrolyte Abnormality Requiring Replacement
Description: Severe electrolyte abnormalities requiring aggressive replacement defined as potassium levels less than 3.0 meq/L during the study.
Time Frame: 48 Hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Placebo | Experimental: Metolazone
Number analyzed (Participants) | 66 | 66
Participants | 0 | 3
Statistical Analysis 1: Comparison: Experimental: Placebo vs Experimental: Metolazone; Test type: Superiority; p = .080, Chi-squared

12. Other Pre Specified Outcome: Number of Participants With Magnesium Electrolyte Abnormality Requiring Replacement
Description: Number of Participants with severe electrolyte abnormalities requiring aggressive replacement defined as magnesium levels less than 1.5 meq/L during the study.
Time Frame: 48 Hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Placebo | Experimental: Metolazone
Number analyzed (Participants) | 66 | 66
Participants | 2 | 1
Statistical Analysis 1: Comparison: Experimental: Placebo vs Experimental: Metolazone; Test type: Superiority; p = .559, Chi-squared

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse effects will be collected for the first 48 hours following enrollment in the MELT trial. No other adverse events are reported unless deemed to related to the study by the Principal Investigator. All cause mortality was assessed and reported for all patients at the 30 day timepoint following study enrollment. Study design did not require collection of mortality data past the 30 day timepoint.
Description: Non-serious adverse effects collected were: Hypotension requiring intervention, electrolyte imbalance requiring intervention and acute kidney injury defined as 30% rise in creatinine over baseline. Per study design All-Cause Mortality, Serious Adverse Events and Non-Serious adverse events reporting include all subjects who received at least one dose of study drug per. Note: Per protocol only patients receiving both doses of study drug were included in primary and secondary measures analysis.
Arm/Group | Experimental: Placebo | Experimental: Metolazone
All-Cause Mortality (participants affected / at risk) | 1/70 | 4/72
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/72
Other Adverse Events (participants affected / at risk) | 13/70 | 15/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Placebo (N=70) | Experimental: Metolazone (N=72)
Hypotension Requiring Intervention (Cardiac disorders) | 6 (6) | 1 (1) — Hypotension Requiring Intervention defined as MAP less than 55
Electrolyte abnormalities requiring intervention (General disorders) | 2 (2) | 4 (4) — Severe electrolyte abnormalities requiring aggressive replacement defined as potassium levels less than 3.0 meq/L or magnesium levels less than 1.5 meq/L during the study.
Acute Kidney Injury (Renal and urinary disorders) | 4 (4) | 10 (10) — Acute kidney injury defined as a 30% rise in creatinine from baseline.
Hypotention requiring intervention and Acute Kidney Injury (General disorders) | 1 (1) | 0 (0) — Hypotention defined as MAP < 50 and AKI defined as 30% increase in creatinine over baseline.

LIMITATIONS AND CAVEATS:
Recruitment ended early due to limited resources,however all protocol directed measures were completed for all enrolled. I&O was measured and recorded manually which introduces room for error.BORG assessment timing not exact due to limited resources.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT02620384/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/84/NCT02620384/SAP_001.pdf